CLINICAL TRIAL: NCT06314139
Title: Tolerability and Efficacy of Continuous Theta-burst Stimulation for Essential Tremor: A Randomized, Double-Blind, Sham-Controlled Study.
Brief Title: Tolerability and Efficacy of Continuous Theta-burst Stimulation for Essential Tremor: A Randomized Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yanming Xu, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YanmingXu001
Record Dates: First submitted 2023-12-05; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Essential Tremor; Continuous Theta Burst Stimulation
Keywords: Essential tremor; Transcranial magnetic stimulation; Continuous theta-burst stimulation; RCT
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cTBS group (Active Comparator): cTBS at 80% action motor threshold (AMT) with 600 pulses over bilateral M1 and cerebellum. Continuous theta-burst stimulation (cTBS) was performed with a CCY-I Magnetic Stimulator (YIRUIDE Medical Co., Wuhan, China) with an air-cooled, figure-of-eight 70 mm coil. The site of stimulation during the TMS treatment sessions was bilateral M1 and cerebellum.
  Interventions: Device: continuous theta-burst stimulation (cTBS)
- sham group (Sham Comparator): Sham stimulation was performed with the same protocol using an inactive coil to mimic true stimulation sound effects, but does not stimulate the brain or produce neurophysiological changes in cerebello-thalamo-cortical (CTC) connections and eyeblink regulation.
  Interventions: Device: continuous theta-burst stimulation (cTBS)

INTERVENTIONS:
Device: continuous theta-burst stimulation (cTBS) — Continuous theta-burst stimulation (cTBS) was performed with a CCY-I Magnetic Stimulator (YIRUIDE Medical Co., Wuhan, China) with an air-cooled, figure-of-eight 70 mm coil. The site of stimulation during the TMS treatment sessions was bilateral M1 and cerebellum. Real cerebellar cTBS was delivered with the coil positioned over the cerebellar hemisphere, i.e., 3 cm laterally to and 1 cm below the inion. The cTBS protocol uses a complex pattern of stimulation consisting of three-pulse bursts at 50 Hz repeated every 200ms. A total of 600 pulses that lasts for about 40 seconds were applied which could result in a sustained reduction in corticospinal excitability that outlasted the period of stimulation by 45 min. It was delivered at an intensity corresponding to 80 % of the active motor threshold (AMT), this is the minimum stimulation intensity that evokes MEPs of approximately 200 μV in amplitude in tonically contracted muscles.

SUMMARY:
Essential tremor (ET) is one of the most common movement disorders in adults. The prevalence rate among the elderly over 65 years old is about 4.6%. Tremor usually worsens with age, leading to disability and loss of independence, which has an adverse impact on the quality of life of patients. However, the traditional first-line treatment drugs are neither effective enough nor completely safe for ET patients. Although surgical procedures such as deep brain stimulation (DBS) and thalamotomy can be used to better control unilateral limb tremor, many patients are reluctant to choose surgical treatment because it's invasive. Therefore, there is an urgent need to develop new drugs or non-invasive therapies as a better treatment option for ET.

The pathology of the disease is not yet clear, it is generally believed that genetic, aging and environmental factors are related to ET. Hyperactivity of cerebellar function and changes of cerebello-thalamo- cortical (CTC) pathways are currently considered to be the most important pathophysiological mechanisms of ET. Therefore, the cerebellum and cortex may be the best targets for the treatment of tremor.

Continuous theta burst stimulation (cTBS) is one of the non-invasive electrophysiological techniques characterized by plexus stimulation, which is similar to low-frequency repetitive transcranial magnetic stimulation (rTMS) but closer to the physiological state of neural activity, and may inhibit the excitability of the stimulated cortex. The stimulation duration is greatly shortened, which is simpler and easier than the low-frequency rTMS of 20-30 minutes. In addition, functional near infrared spectroscopy (fNIRS) is a new non-invasive functional neuroimaging technique. It mainly uses the difference characteristics of oxyhemoglobin and deoxyhemoglobin in brain tissue for near-infrared light absorption at different wavelengths of 600-900nm. The efficacy, safety, and mechanisms involved in non-invasive stimulation therapy for ET patients are still unclear. There are few studies on the treatment of ET with cTBS, and the sample size is small (the largest sample includes only 23 ET patients). Additionally, there was a lack of exploration on the therapeutic mechanism of cTBS for ET patients. Therefore, the investigators conducted a double-blind, randomized, sham-controlled clinical trial to evaluate the safety and efficacy of cTBS in the treatment of ET patients over both cerebellar and cortical area.

DETAILED DESCRIPTION:
Essential tremor (ET), also known as idiopathic tremor, is one of the most common movement disorders in adults. The prevalence rate among the elderly over 65 years old is about 4.6%. It is characterized by simple kinetic and/or postural tremor of the arms, with or without various combinations of midline tremors (MT)-such as the neck, voice, and facial tremors. About 30%~70% of ET patients have family history, and most of them are autosomal dominant. Tremor usually worsens with age, leading to disability and loss of independence, which has an adverse impact on the quality of life of patients. However, the traditional first-line treatment drugs are neither effective enough nor completely safe for ET patients. Although surgical procedures such as deep brain stimulation (DBS) and thalamotomy can be used to better control unilateral limb tremor, many patients are reluctant to choose surgical treatment because it's invasive. Therefore, there is an urgent need to develop new drugs or non-invasive therapies as a better treatment option for ET.

The pathology of the disease is not yet clear, it is generally believed that genetic, aging and environmental factors are related to ET. Hyperactivity of cerebellar function and changes of cerebello-thalamo- cortical (CTC) pathways are currently considered to be the most important pathophysiological mechanisms of ET. The degenerative changes of cerebellum in ET patients are prominent, such as the loss of Purkinje cells and focal axonal swelling. In addition, imaging, electrophysiological studies and clinical observations show that the cerebral cortex may also be involved. Studies have shown that the activity of cortical area is related to the frequency of tremor, and there have been reports on the disappearance of ET after cortical infarction. Therefore, the cerebellum and cortex may be the best targets for the treatment of tremor.

Transcranial magnetic stimulation (TMS) is a non-invasive electrophysiological technique for nerve stimulation and nerve regulation invented by Anthony Barker in 1985. Its principle is to use electromagnetic fields to generate induced electric fields in the brain, change abnormal brain waves of patients, and regulate the secretion of neurotransmitters and hormones closely related to emotion, cognition, sleep and other functions in the brain, so as to achieve the therapeutic effect. Continuous theta burst stimulation (cTBS) is characterized by plexus stimulation, which is similar to low-frequency rTMS but closer to the physiological state of neural activity, and may inhibit the excitability of the stimulated cortex. Moreover, the intervention time of CTBS is only 40 seconds, the stimulation intensity is lower, and the stimulation duration is greatly shortened, which is simpler and easier than the low-frequency rTMS of 20-30 minutes. The investigators hypothesized that CTBS would reduce the excitability of cerebellar cortex, thereby reducing the amplitude of tremor, and play a therapeutic role in ET patients.

Functional near infrared spectroscopy (fNIRS) is a new non-invasive functional neuroimaging technique in recent years. fNIRS mainly uses the difference characteristics of oxyhemoglobin and deoxyhemoglobin in brain tissue for near-infrared light absorption at different wavelengths of 600-900nm to directly detect the hemodynamic activities of cerebral cortex in real time, and then through observing such hemodynamic changes, discover the neurovascular coupling law, so as to deduce the neural activities of the brain. In the past 20 years, the hardware manufacturing and improvement of functional near-infrared spectroscopy technology and data processing methods have become more and more perfect, making the fNIRS technology, which uses near-infrared light to observe brain neural activities, to study various cognitive activities emerge in endlessly and develop rapidly. fNIRS is based on light intensity. Optical imaging equipment has high cost performance and is not vulnerable to electromagnetic interference from TMS pulses. It can conduct more detailed research on cortical connectivity, excitability and dynamic changes induced by cTBS.

Studies by Chuang et al. showed that after the treatment of cTBS over motor cortex or premotor cortex, the tremor amplitude of ET patients decreased significantly, but the tremor frequency remained unchanged. Hellriegel et al. included 10 ET patients and 10 healthy controls. They performed a single cTBS treatment on the primary motor cortex of the patients. They found that compared with the control group, the cTBS group reduced the total power of tremor assessed by the accelerometer, but this beneficial effect was subclinical, that is, the tremor assessment of the patients had no significant change before and after treatment. Bologna et al. included 16 ET patients and 11 healthy controls. They were treated with cTBS and sham stimulation in the right cerebellar hemisphere with crossing over after a one-week washout period. The results showed that the tremor was not significantly improved before and after CTBS treatment. They also pointed out that multiple stimuli may be effective. However, there is a lack of research on the therapeutic mechanism of cTBS in the treatment of ET. The combination of transcranial magnetic stimulation (TMS) and neuroimaging provides a new way to explore the mechanisms involved. High frequency rTMS could improve mild cognitive impairment after stroke and increase the concentration of oxyhemoglobin in prefrontal lobe. Study have observed the changes of activation mode of cerebral cortex during upper limb movement in stroke patients before and after repeated transcranial magnetic stimulation (rTMS) treatment through near infrared brain functional imaging (fNIRS). Struckmann et al. used fNIRS technology to compare the changes of prefrontal blood oxygen response in patients with depression before and after intermittent TBS treatment. They also confirmed that the oxygen and hemoglobin of patients did change before and after treatment, and further discussed the mechanism.

To sum up, there are few domestic and international clinical studies on the treatment of ET with CTBS, and the sample size is small (the largest sample includes only 23 ET patients). The results showed that the placebo effect was strong, and all of them were stimulated by single site, and the effect was not significant. Additionally, there was a lack of exploration on the therapeutic mechanism of cTBS for ET patients. Therefore, The investigators will conduct a double-blind, randomized, sham-controlled clinical trial to evaluate the safety and efficacy of cTBS in the treatment of ET patients over both cerebellar and cortical area. fNIRS technology will be applied to provide new ideas for the pathophysiological mechanism and treatment of ET.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Right-hand dominant
* Were willing to participate in the trial and signed informed consent
* Essential tremor Diagnosis based on the International Parkinson and Movement Disorder Society (IPMDS) ET diagnostic criteria in 2017

Exclusion Criteria:

* A history of trauma 3 months before the onset of the disease, and it can be clearly determined that this history of trauma has led to neurological dysfunction
* Combined with other central nervous system diseases except ET
* drug or alcohol withdrawal-induced tremor, psychogenic/physiological/orthostatic/task-specific tremor
* Contraindications for undergoing cTBS, such as epilepsy history, intracranial metal implants, pacemaker installers, etc
* Skin lesions at stimulation sites
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Tremor assessment using Fahn-Tolosa-Marin (FTM) tremor-rating scales | All participants were assessed at baseline, 0 minutes, 10 minutes and 45 minutes post-intervention.
  The primary outcome was tremor assessment using Fahn-Tolosa-Marin tremor-rating scales (FTMTRS). All participants were assessed at baseline, 0 minutes, 10 minutes and 45 minutes post-intervention. Clinical assessment was independently performed by a neurologist specialized in movement disorder, using the Fahn-Tolosa-Marin (FTM) tremor-rating scales which comprises parts A, B and C, to evaluate severity and forms of tremor symptoms. (tremor severity: part A, specific writing/drawing tasks: part B, and functional disability: part C). Each item has 5 levels of scores (0, 1, 2, 3, and 4), representing different degrees of tremor in the patient. The total score of FTMTRS ranges from 0 to 160. The higher the score, the more severe the tremor.

SECONDARY OUTCOMES:
Clinical global impression-improvement (CGI-I) rating scores | Clinical global impression-improvement (CGI-I) rating scores were assessed approximately 45 minutes after intervention.
  The secondary outcome 2 was the clinical global impression-improvement (CGI-I) rating score. The CGI-I rating scale is composed of the following three parts: severity of illness (SI), global improvement (GI) and efficacy index (EI), which are used to evaluate the clinical efficacy of treatment. The severity of the disease (SI) is compared with other patients in the same study to assess the current condition of the subjects. The global improvement (GI) is to assess whether there is any change in the current condition of the evaluated patients relative to their baseline state prior to the study. Both SI and GI are scored at 8 levels of 0-7. The efficacy index comprehensively considers the efficacy and side effects of the study treatment itself, and its total score range is 0~4.0.
Electrophysiological evaluation of cortical excitability and inhibition measured by TMS. | Electrophysiological evaluation of cortical excitability and inhibition by transcranial magnetic stimulation (TMS) were assessed at baseline and approximately 45 minutes after intervention.
  The secondary outcome 3 was electrophysiological evaluation of cortical excitability and inhibition measured by transcranial magnetic stimulation. Electrophysiological parameters include rest motor threshold (RMT), intracortical inhibition (ICI) with stimulation interval of 1ms and 2ms, intracortical facilitation (ICF) with stimulation interval of 12ms and 15ms, and cortical silent period (CSP).

CONTACTS AND LOCATIONS:
Overall Officials: Xu Yanming, Study Director — Department of Neurology, West China Hospital, Sichuan University
Locations (1):
- Department of Neurology, West China Hospital, Sichuan University, 37 Guo Xue Xiang, Chengdu, Sichuan Province 610041, P.R. China., Chengdu, Sichuan, China